CLINICAL TRIAL: NCT01560481
Title: Randomized Clinical Trial to Evaluate Safety, Tolerability and PK-PD Profile of Metformin Glycinate 620 mg,1240 mg, 2480 mg and Metformin Chlorhydrate 1000 mg of One Single Dose, Multiple Dose and After Food Intake.
Brief Title: Clinical Trial to Evaluate Safety and pK Profile of Metformin Glycinate in Healthy Volunteers
Acronym: NTC00940472
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NTC00940472
Record Dates: First submitted 2012-02-09; First posted 2012-03-22 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: metformin glycinate; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — Eating; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Step A: metformin glycinate 620 mg (Experimental): 620mg single dose by mouth
  Interventions: Drug: Step A: metformin glycinate 620 mg single dose
- Step A: metformin glycinate 1240 mg (Experimental): 1240mg single dose by mouth
  Interventions: Drug: Step A: metformin glycinate 1240 mg single dose
- Step A: metformin glycinate 2480 mg (Experimental): 2480mg single dose by mouth
  Interventions: Drug: Step A: metformin glycinate 2480 mg single dose
- Step A: metformin hydrochloride 1000 mg (Active Comparator): 1000mg single dose by mouth
  Interventions: Drug: Step A: metformin hydrochloride 1000 mg single dose
- Step A: metformin glycinate 1240 mg, food intake (Experimental): 1240mg single dose by mouth after food intake
  Interventions: Drug: Step A: metformin glycinate 1240 mg,food intake
- Step B: metformin glycinate 620 mg BID (Experimental): 620mg BID for 8 days
  Interventions: Drug: Step B: metformin glycinate 620 mg BID
- Step B: metformin hydrochloride 500 mg BID (Active Comparator): 500mg tablets BID for 8 days
  Interventions: Drug: Step B: metformin hydrochloride 500 mg BID

INTERVENTIONS:
Drug: Step A: metformin glycinate 620 mg single dose — metformin glycinate 620 mg single dose
  Arms: Step A: metformin glycinate 620 mg
Drug: Step A: metformin glycinate 1240 mg single dose — metformin glycinate 1240 mg single dose
  Arms: Step A: metformin glycinate 1240 mg
Drug: Step A: metformin glycinate 2480 mg single dose — metformin glycinate 2480 mg single dose
  Arms: Step A: metformin glycinate 2480 mg
Drug: Step A: metformin hydrochloride 1000 mg single dose — metformin Chlorhydrate 1000 mg single dose
  Arms: Step A: metformin hydrochloride 1000 mg
Drug: Step A: metformin glycinate 1240 mg,food intake — metformin glycinate 1240 mg, intake of food
  Arms: Step A: metformin glycinate 1240 mg, food intake
Drug: Step B: metformin glycinate 620 mg BID — metformin glycinate 620 mg BID, 8 days
  Arms: Step B: metformin glycinate 620 mg BID
Drug: Step B: metformin hydrochloride 500 mg BID — metformin Chlorhydrate 500 mg BID, 8 days
  Arms: Step B: metformin hydrochloride 500 mg BID

SUMMARY:
Metformin Glycinate is a novel biguanide compound developed as a potential candidate for the treatment of type 2 diabetes. Metformin Glycinate was found to improve metabolic control in naive patients with type 2 diabetes.

The objective of this study is to evaluate the safety, tolerability and pK profile of Metformin Glycinate 620 mg QD, 1240 mg QD, 2480 mg QD, after administration of one single dose, in step A. In step A will be included 25 volunteers.

In step B the objective is to evaluate Safety, tolerability and pK profile of Metformin Glycinate 620 mg BID, after administration of multiple dose during 8 days. In step B will be included 24 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years.
* Weight within normal ranges (Quetelet index between 21 and 26) (weight (kg)/height (m2).
* Adequate physical examination and clinical history
* No organic and psychiatric disorder
* Normal Blood pressure, Pulse Rate, temperature and ECG.
* Lab test within normal values according to reference lab values of Biochemistry lab of Hospital Santa Creu I Sant Pau. It will be allowed changes according to clinical criteria of the clinical staff of ICIM-SANT PAU
* Females of childbearing potential with adequate contraceptive precautions, other than oral contraceptives and negative urine pregnancy test.
* No participation in any other clinical trial within the previous two months before the initiation of this study.
* No blood donation within the previous four weeks before the initiation of this study.
* Signed informed consent.

Exclusion Criteria:

* Drugs or alcohol abuse.
* Consumer of stimulant drinks (> 5 coffees, teas, cola drinks).
* Smokers (> 10 cigars).
* Precedents of drugs allergy or hypersensitivity
* Intake of any other medication within the previous 15 days before this study.
* Positive HIV, HBV or HCV.
* Chronic disease (cardiovascular, respiratory, endocrine, gastrointestinal, hematologic, neurologic or others).
* Prior surgery within the previous six months before the initiation of this study.
* Pregnant women or breastfeeding or females of childbearing potential with no adequate contraceptive precautions, other than oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Step A: Number of Adverse Events of Metformin Glycinate 620 mg QD, 1240 mg QD, 2480 mg QD, after administration of one single dose | 35 days
  Tolerability:
  * adverse events,
  * systolic and diastolic blood pressure, pulse rate and temperature
  * pulse rate and ECG alterations
  * alterations in haematology, plasma chemistry, and urine analyses
Step B: Number of Adverse Events of Metformin Glycinate 620 mg BID, after administration of multiple dose during 8 days | 25 days
  Tolerability:
  * adverse events,
  * systolic and diastolic blood pressure, pulse rate and temperature
  * pulse rate and ECG alterations
  * alterations in haematology, plasma chemistry, and urine analyses

SECONDARY OUTCOMES:
Step A: Bioavailability (AUC) of metformin glycinate 620 mg QD, 1240 mg QD, 2480 mg QD after administration of one single dose with metformin Chlorhydrate 1000 mg QD. | 36 hours
Step A: Linear and dose-proportional (AUC) pharmacokinetic of 620 mg, 1240 mg and 2480 strengths of metformin glycinate | 36 hours
Step A: Bioavailability (AUC) of metformin glycinate 1240 mg QD in fasted subjects and after the intake of fat rich breakfast | 36 hours
Step A: Pharmacokinetic profile (AUC) of metformin glycinate 620mg QD, 1240 mg QD, 2480 mg QD after administration one single dose and pharmacokinetic profile of metformin chlorhydrate 1000mg QD. | 36 hours
Step B: Bioavailability (AUC) of metformin glycinate 620 mg BID and bioavailability of metformin chlorhydrate 500mg BID, after administration of multiple doses during 8 days. | 8 days
Step B: Pharmacokinetic profile (AUC) of metformin glycinate 620mg BID after administration of multiple doses during 8 days | 8 days
Step A: Bioavailability (Cmax) of metformin glycinate 620 mg QD, 1240 mg QD, 2480 mg QD after administration of one single dose with metformin Chlorhydrate 1000 mg QD. | 36 hours
Step A: Linear and dose-proportional pharmacokinetic (Cmax) of 620 mg, 1240 mg and 2480 strengths of metformin glycinate | 36 hours
Step A: Bioavailability (Cmax) of metformin glycinate 1240 mg QD in fasted subjects and after the intake of fat rich breakfast | 36 hours
Step A: Pharmacokinetic profile (Cmax) of metformin glycinate 620mg QD, 1240 mg QD, 2480 mg QD after administration one single dose and pharmacokinetic profile of metformin chlorhydrate 1000mg QD. | 36 hours
Step B: Bioavailability (Cmax) of metformin glycinate 620 mg BID and bioavailability of metformin chlorhydrate 500mg BID, after administration of multiple doses during 8 days. | 8 days
Step B: Pharmacokinetic profile (Cmax) of metformin glycinate 620mg BID after administration of multiple doses during 8 days | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Antonijoan, MD, Study Chair — Centre d'Investigació de Medicaments Hospital de la Santa Creu i Sant Pau
Locations (1):
- Centre d'Investigació de Medicaments Hospital de la Santa Creu i Sant Pau, Barcelona, Spain